CLINICAL TRIAL: NCT01293500
Title: Goal-directed Resuscitative Interventions During Pediatric Inter-facility Transport (The GRIPIT Trial)
Acronym: GRIPIT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1R21HD060171-01A2 (NIH)
Record Dates: First submitted 2010-10-22; First posted 2011-02-10 (Estimated); Last update posted 2025-10-02 (Actual); Status verified 2016-05

CONDITIONS: Systemic Inflammatory Response Syndrome
Keywords: SIRS; shock; sepsis; pediatric; inter-facility transport; specialized transport; NIRS monitoring
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome; Shock; Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Goal-directed Therapeutic Protocol — A 10 month period of data collection for transport patients with SIRS (Systemic Inflammatory Response Syndrome) will be followed by training and institution of a goal-directed resuscitation protocol. A second 10 month data collection period will then commence. Groups will be compared with respect to outcome measures at the end of the study. All subjects will be monitored with NIRS cerebral and somatic oximetry.

SUMMARY:
Recent advances in critical care medicine have dramatically improved morbidity and mortality of critical illness. Goal-directed therapy protocols have been instrumental in this change. Goal-directed therapy standardizes the rapid delivery of definitive care in illnesses such as SIRS (Systemic Inflammatory Response Syndrome) and head trauma. Although this treatment approach has been shown to improve clinical outcomes, it has not been widely adopted outside academic medical centers. Further improvement in outcomes of critical illness is likely if goal-directed therapy is utilized early in the course of care. To facilitate this early adoption, goal-directed therapeutic protocols should be developed and implemented by specialized pediatric transport teams. The investigators hypothesize that the institution of goal-directed therapy during pediatric interfacility transport will improve the outcomes of critically ill children.

The GRIPIT Trial (Goal-directed Resuscitative Interventions during Pediatric Inter-facility Transport) will compare outcomes of pediatric SIRS patients before and after the implementation of a goal-directed therapeutic protocol during transport. This will be the first test of goal-directed therapy in the transport environment. Data will be collected on pediatric SIRS patients transported by the Angel One Transport Team at Arkansas Children's Hospital before and after protocol implementation. Outcome measures will include length of hospital stay, length of intensive care unit (ICU) stay, incidence of multiple organ dysfunction syndrome (MODS), and required therapeutic interventions during ICU stay (TISS-28 scores). In addition, NIRS (Near-Infrared Spectroscopy) monitoring will be used as a cerebral and somatic oxygenation trend monitor, to determine its effectiveness as a resuscitation guide for pediatric SIRS during transport. NIRS trends are useful as a surrogate marker for systemic venous saturations, known to decrease with severe SIRS.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients transported to Arkansas Children's Hospital by the Angel One Transport Team
* Age Group: 1 month - 17 years
* Systemic Inflammatory Response Syndrome (Age-specific SIRS criteria)

Exclusion Criteria:

* Known or suspected congenital heart disease
* Known or suspected cardiomyopathy or myocarditis
* Diabetic Ketoacidosis (DKA) as SIRS-inducing illness
* Traumatic Brain Injury (TBI) as SIRS-inducing illness
* Burn Injury as SIRS-inducing illness
* Patients with known or suspected active hemorrhage

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 230 (Actual)
Dates: Start 2010-10; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Incidence of Multiple Organ Dysfunction | ICU Admission to ICU Discharge
  Computed utilizing PELOD scores.
Required ICU Interventions | ICU Admission to ICU Discharge
  Utilizing TISS-28 Scores
Hospital Length of Stay | Hospital Admission to Hospital Discharge
  Subjects will be followed from hospital admission to hospital discharge.

SECONDARY OUTCOMES:
Changes in cerebral and somatic oxygenation | During Inter-facility Transport (Average)
  Utilizing NIRS Technology

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Stroud, MD, Principal Investigator — Arkansas Children's Hospital Research Institute
Locations (1):
- Arkansas Children's Hospital, Little Rock, Arkansas, United States

REFERENCES:
- [Derived] Stroud MH, Sanders RC Jr, Moss MM, Sullivan JE, Prodhan P, Melguizo-Castro M, Nick T. Goal-Directed Resuscitative Interventions During Pediatric Interfacility Transport. Crit Care Med. 2015 Aug;43(8):1692-8. doi: 10.1097/CCM.0000000000001021. PMID 25860203